CLINICAL TRIAL: NCT06048484
Title: A Phase 2, Open-Label, Multicenter, Randomized Study Evaluating Neoadjuvant Therapy Targeting the Adenosine Immunosuppressive Pathway in Combination With Immune Checkpoint Blockade and Radiation Therapy in Patients With Advanced PANCreatic Ductal Adenocarcinoma Who Are Candidates for Surgical Resection
Brief Title: Combination Therapy in Patients With Localized Pancreatic Ductal Adenocarcinoma
Acronym: AIRPanc
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gulam Manji (Other)
Collaborators: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Gulam Manji, Associate Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAU4206
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Radiosurgery; zimberelimab; quemliclustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: Safety run-in (Experimental): Prior to resection: SBRT 40 Gy over 5 fractions, zimberelimab (AB122) 240 mg intravenously (IV) every 2 weeks for 7 weeks (4 doses), quemliclustat (AB680) 100 mg IV every 2 weeks for 7 weeks (4 doses) and etrumadenant (AB928) 150 mg PO daily for 7 weeks. After resection: mFOLFIRINOX (4 cycles)
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT); Drug: Zimberelimab; Drug: Quemliclustat; Drug: Etrumadenant; Drug: Modified FOLFIRINOX
- Arm B: SBRT with Zimberelimab (AB122) Alone (Control Arm) (Active Comparator): Prior to resection: SBRT 40 Gy over 5 fractions, 240 mg IV zimberelimab (AB122) every 2 weeks for 7 weeks (4 doses) prior to surgery. After resection: mFOLFIRINOX (4 cycles)
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT); Drug: Zimberelimab; Drug: Modified FOLFIRINOX
- Arm C: SBRT, Zimberelimab with quemliclustat (AB680) (Experimental): Prior to resection: SBRT 40 Gy over 5 fractions, 240 mg IV zimberelimab (AB122) every 2 weeks for 7 weeks (4 doses) prior to surgery in combination with quemliclustat IV at the recommended therapeutic dose (RTD)every 2 weeks for 7 weeks (4 doses) prior to surgery. After resection: mFOLFIRINOX (4 cycles)
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT); Drug: Zimberelimab; Drug: Quemliclustat; Drug: Modified FOLFIRINOX
- Arm D: SBRT, Zimberelimab with AB680 and Etrumadenant (AB928) (Experimental): Prior to resection: SBRT 40 Gy over 5 fractions, 240 mg IV zimberelimab (AB122) every 2 weeks for 7 weeks (4 doses) prior to surgery in combination with quemliclustat IV at the RTD every 2 weeks for 7 weeks (4 doses) and etrumadenant (AB928) PO at the RTD daily for 7 weeks prior to surgery. After resection: mFOLFIRINOX (4 cycles)
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT); Drug: Zimberelimab; Drug: Quemliclustat; Drug: Etrumadenant; Drug: Modified FOLFIRINOX

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy (SBRT) — SBRT 40 gray (Gy) over 5 fractions
Drug: Zimberelimab — 240 mg intravenously (IV)
  Other Names: AB122
Drug: Quemliclustat — 100 mg IV
  Other Names: AB680
  Arms: Arm A: Safety run-in; Arm C: SBRT, Zimberelimab with quemliclustat (AB680); Arm D: SBRT, Zimberelimab with AB680 and Etrumadenant (AB928)
Drug: Etrumadenant — 150 mg orally
  Other Names: AB928
  Arms: Arm A: Safety run-in; Arm D: SBRT, Zimberelimab with AB680 and Etrumadenant (AB928)
Drug: Modified FOLFIRINOX — * Oxaliplatin 85 mg per square meter IV
  * Irinotecan 150 mg per square meter IV
  * Leucovorin 400 mg per square meter IV
  * Fluorouracil 2400 mg per square meter IV
  * Pegfilgrastim injector kit (6mg subcutaneous)
  Other Names: mFOLFIRINOX

SUMMARY:
The purpose of this study is to combine standard radiation therapy with drugs that encourages the body's immune system against cancer cells and simultaneously adding drugs which also target the pathway that the tumor uses to evade the immune system (CD73 and A2a/b). The study hopes that these drugs will work in concert with radiation therapy to kill cancer cells.

The specific goal of this study is to ensure that treatment with zimberelimab and stereotactic body radiation therapy (SBRT) alone or in combination with quemliclustat (a drug which blocks CD73), with or without etrumadenant (a drug which blocks the A2a/b) given before surgery is safe and if it can further increase the immune response against the tumor.

DETAILED DESCRIPTION:
The overall objective of this study is to combine standard radiation therapy with drugs that stimulate the body's immune system against cancer cells (by targeting the protein programmed cell death (PD-1), while adding drugs which also target the pathway that the tumor uses to evade the immune system (the CD73 and A2a/b pathways).The main goal of this study is to find out if study treatment with zimberelimab (an antibody which binds the protein PD-1) and stereotactic body radiation therapy (SBRT) alone or in combination with quemliclustat (a drug which blocks CD73), with or without etrumadenant (a drug which blocks the A2a/b) given before surgery is safe and if it can further increase the immune response against the tumor.

The study is divided into two parts (Stage 1 and Stage 2). In Stage 1 participants will undergo 5 days of SBRT and receive zimberelimab, quemliclustat and etrumadenant (Arm A) for 7 weeks before surgery. If this combination is considered safe, the study will proceed to Stage 2. In Stage 2, participants will be randomized into one of three different treatment arms (B - D). All participants will undergo SBRT and will receive either Zimberelimab alone (Arm B), a combination of zimberelimab with quemliclustat (Arm C), or will receive combination of zimberelimab, quemliclustat and etrumadenant (Arm D) for 7 weeks prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histological or pathological confirmation of pancreatic adenocarcinoma Cytologic or histologic proof of pancreatic ductal adenocarcinoma (PDAC) needs to be verified by the treating institution pathologist. A pathological report from non-treating institutions is sufficient to consent and to initiate investigational therapy if tissue sample is unavailable for evaluation at time of consent or enrollment. However, in such a case, PDAC diagnosis should be confirmed by the treating institution pathologist at a later time.
* Completed 8 cycles of neoadjuvant modified FOLFIRINOX. Omission of oxaliplatin due to adverse events may be allowed in cycles 5-8 with consultation with the principal investigator.
* Patients with surgically resectable PDAC who are considered appropriate to undergo the applicable operation.
* Eligible to undergo SBRT.
* Measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* No prior surgical, systemic, or radiotherapy for PDAC except for mFOLFIRINOX.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Age ≥ 18 years.
* Adequate hematological and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of investigational treatment:

Exclusion Criteria:

* Prior treatment with T-cell co-stimulating or immune checkpoint blockade therapies, including but not limited to anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies.
* Patients who are receiving any other investigational agents concurrently.
* Concomitant treatment with other anti-neoplastic agents (hormonal therapy acceptable).
* Uncontrolled pleural effusion, pericardial effusion, or ascites.
* Uncontrolled hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL, or corrected serum calcium > ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy.
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease (Crohn's disease or ulcerative colitis), antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis (some exceptions permissible as outlined per protocol).
* History of idiopathic pulmonary fibrosis, interstitial lung disease, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.

  • History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Positive HIV test at screening or at any time prior to screening.
* Active hepatitis B virus (HBV) infection (chronic or acute), defined as having a positive hepatitis B surface antigen (HBsAg) test at screening.

  --Note: Patients with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total hepatitis B core antibody test at screening, are eligible for the study.
* Active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test followed by a positive HCV RNA test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
* Known clinically significant liver disease, including alcoholic hepatitis, cirrhosis, fatty liver disease, and inherited liver disease.
* Known active tuberculosis.
* Inability to swallow medication or malabsorption condition that would alter the absorption of orally administered medications.
* Pregnant women are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents and breastfeeding should be discontinued.
* History of allergy or hypersensitivity to oxaliplatin, irinotecan, leucovorin, fluorouracil, pegfilgrastim, or any excipients.
* History of Gilbert's disease or known genotype UGT1A1 *28/*28.
* Inflammatory disease of the colon or rectum, or severe uncontrolled diarrhea.
* Active or history of celiac disease.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in the number of intratumoral CD8+ T-cells | Perioperative
  The primary endpoint is change in the number of intratumoral CD8+ T-cells at time of surgery between treatment arm(s) compared to the SBRT + zimberelimab arm (Control Arm B). To obtain CD8+ T-cell count, simple immunohistochemistry (IHC) will be used to quantitate CD8+ T-cells. A designated gastrointestinal (GI) pathologist will review each hematoxylin and eosin (H&E) stained serial section and IHC slide to oversee the process. Representative areas within the slide will be used for cell counts.

SECONDARY OUTCOMES:
Resection rate | Week 8
  The proportion of patients undergoing surgical resection after randomization. Patients that do not undergo an explorative laparotomy at all or do undergo an explorative laparotomy but not a resection are considered a failure.
Microscopically Negative Margins (R0) resection rate | Week 8
  R0 resection rate: Defined as the percentage of eligible patients who underwent surgery with microscopically negative margins (R0). The resection is considered R0 if the inked margin is further than 1 mm distinct from any tumor cells.
  .
Pathologic Complete Response Rate | Week 8
  Pathologic complete response rates after R0 or R1 resection as per the Modified Ryan Scheme for Tumor Regression Score (no viable cancer cells). R0 defined as inked margin is further than 1 mm distinct from any tumor cells. R1 defined as macroscopically curative resection, but tumor cells are observed by microscopy at one or more edges of the resected specimen.
Recurrence free survival | 18 months
  Defined as investigator assessed survival without overt recurrent pancreatic cancer from the date of randomization. Any sign of recurrent or persistent disease, locoregional or distant, as well as death from any cause is considered an event for this endpoint. Recurrence of disease is defined as radiological evidence of recurrence that is confirmed by biopsy. However, if recurrence is suspected due to participant symptoms consistent with disease recurrence and rising tumor markers (that are not explained due to inflammation or biliary obstruction) may result in sooner scans. All efforts will be made to confirm recurrence by conducting a biopsy if considered safe. If a patient is unable to undergo biopsy to confirm recurrence, these cases will be discussed at the institutional multidisciplinary conference for consensus and discussed with the overall study principal investigator (PI) and the participant will be deemed to have clinical recurrence.
Overall Survival | 4 years
  Defined as the period of time between randomization and death from any cause. Participants alive at last follow-up are censored.
Count of Grade 3 or Higher Adverse Events | 4 months
  The safety profile will be assessed by the count of grade 3 or higher adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Gulam Manji, MD, PhD, Principal Investigator — Columbia University
Locations (5):
- United States (5):
  - Northwell Health R.J. Zuckerberg Cancer Center, Lake Success, New York
  - Columbia University Irving Medical Center, New York, New York
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin